CLINICAL TRIAL: NCT03217045
Title: Impact of Introducing a Standardized Nutrition Protocol on Very Premature Infants' Growth and Morbidity
Brief Title: Nutrition Protocol and Premature Infants' Growth
Acronym: Nutriproto
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: R2015-1
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Premature Infants; Nutrition Deficiency Due to Insufficient Food; Growth Retardation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before Protocol: 72 premature infants born between 26 and 32 weeks gestation, over 6 months period, and involved before the introduction of a strict nutrition protocol
  Interventions: Other: nutrition protocol introduction
- After Protocol: 86 premature infants born between 26 and 32 weeks gestation, over 6 months period, and involved after the introduction of a strict nutrition protocol and a washout period of 6 months
  Interventions: Other: nutrition protocol introduction

INTERVENTIONS:
Other: nutrition protocol introduction — Growth comparison of 2 cohorts of infants evaluated in a before-after design

SUMMARY:
Nutrition is a major issue for premature infants. Inappropriate nutritional intake during the first weeks of life is responsible for postnatal growth restriction and adverse long-term outcomes.

This study aimed at evaluating the impact of the introduction of an updated, standardized, nutrition protocol on very premature infants' growth and morbidity, and the care givers' compliance to the new protocol.

ELIGIBILITY:
Inclusion Criteria:

* All surviving infants born between 26 and 32 weeks gestation in our Level III NICU

Exclusion Criteria:

* Death
* Any congenital malformation

Ages: 1 Day to 77 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants born between 26 to 32 weeks gestation and admitted to our level III NICU were eligible and included in the study
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
weight | weekly recording from Day 0 up to Day 77
  longitudinal weight evaluation

SECONDARY OUTCOMES:
Necrotizing enterocolitis | Day 77 postnatal age
  Necrotizing enterocolitis
late onset sepsis | Day 77 postnatal age
  Incidence of late onset sepsis
patent ductus arteriosus | Day 77 postnatal age
  Incidence of patent ductus aretriosus requiring treatment
Bronchopulmonary dysplasia | Day 77 postnatal age
  Incidence of Bronchopulmonary dysplasia
Central venous catheters. | Day 77 postnatal age
  Duration of central venous catheters
Compliance to the protocol | weekly recording from Day 0 up to Day 77
  comparison between expected prescription and actual nutrition intake

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wittwer A, Hascoet JM. Impact of introducing a standardized nutrition protocol on very premature infants' growth and morbidity. PLoS One. 2020 May 21;15(5):e0232659. doi: 10.1371/journal.pone.0232659. eCollection 2020. PMID 32437423